CLINICAL TRIAL: NCT01609309
Title: Multicenter Study on Comparison of Long-term Outcome Between Laparoscopic and Open Distal Subtotal Gastrectomy With D2 Lymphadenectomy for Locally Advanced Gastric Cancer
Brief Title: Multicenter Study on Laparoscopic Distal Subtotal Gastrectomy for Advanced Gastric Cancer (CLASS-01)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Guoxin Li, M.D., Ph.D., Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLASS - 01
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms; Laparoscopy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic gastrectomy (Experimental): Laparoscopic distal subtotal gastrectomy with D2 lymphadenectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Laparoscopic gastrectomy
- Open gastrectomy (Active Comparator): Open distal subtotal gastrectomy with D2 lymphadenectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Open gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic gastrectomy — * After exclusion of T4b, bulky lymph nodes, or distant metastasis case by diagnostic laparoscopy, laparoscopic distal subtotal gastrectomy and D2 lymph node dissection will be performed with curative treated intent.
  * The type of reconstruction will be selected according to the surgeon's experience and anastomotic procedure is performed extracorporeally using a mini-laparotomy.
  Other Names: LDG
  Arms: Laparoscopic gastrectomy
Procedure: Open gastrectomy — * After exclusion of T4b, bulky lymph nodes, or distant metastasis case by diagnostic laparoscopy, open distal subtotal gastrectomy and D2 lymph node dissection will be performed with curative treated intent.
  * The type of reconstruction will be selected according to the surgeon's experience.
  Other Names: ODG
  Arms: Open gastrectomy

SUMMARY:
* Laparoscopic distal subtotal gastrectomy with lymph node dissection as minimally invasive surgery has gained popularity for the treatment of early gastric cancer in East Asian countries, even though the long-term follow-up outcome based on multicenter randomized clinical trial (RCT) is still awaited.
* For the patient with locally advanced gastric cancer, several studies indicated that laparoscopic distal subtotal gastrectomy with D2 lymphadenectomy is a technically feasible and safe procedure by experienced surgeons in high-volume specialized hospitals. However, the application of it is controversial mainly due to lack of solid evidence on the oncologic efficacy. Therefore, conventional open approach is still the current standard for advanced gastric cancer.
* Nowadays, the proportion of patients with locally advanced gastric cancer is estimated up to 80 per cent of all gastric cancer cases in China. Before the clinical application of laparoscopic procedure for the treatment with curative intent to advanced gastric cancer located at the middle- or lower-third of the stomach, the oncologic efficacy must be verified.
* Accordingly,the comparison of intraoperative and postoperative complications between laparoscopic and open distal subtotal gastrectomy for over 65 years old patients with gastric cancer based on a randomized controlled trial is needed.

ELIGIBILITY:
Inclusion Criteria:

* Age from over 18 to under 75 years
* Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
* cT2-4a, N0-3, M0 at preoperative evaluation according to the AJCC Cancer Staging Manual Seventh Edition
* Expected curative resection through distal subtotal gastrectomy with D2 lymphadenectomy
* Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale
* ASA (American Society of Anesthesiology) score class I, II, or III
* Written informed consent

Exclusion Criteria:

* Women during pregnancy or breast-feeding
* Severe mental disorder
* History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
* History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection
* Enlarged or bulky regional lymph node diameter over 3cm by preoperative imaging
* History of other malignant disease within past five years
* History of previous neoadjuvant chemotherapy or radiotherapy
* History of unstable angina or myocardial infarction within past six months
* History of cerebrovascular accident within past six months
* History of continuous systematic administration of corticosteroids within one month
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
* FEV1<50% of predicted values

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1056 (Estimated)
Dates: Start 2012-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 36 months

SECONDARY OUTCOMES:
Morbidity and mortality | 30 days; 36 months
  The early postoperative complication and mortality are defined as the event observed within 30 days after surgery, while the time frame for late complication is the period from postoperative day 31th to the end of month 36th.
3-year overall survival rate | 36 months
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type.
Postoperative recovery course | 10 days
  * Time to first ambulation, flatus, liquid diet, soft diet, and duration of hospital stay are used to assess the postoperative recovery course.
  * The amount of abdominal drainage and blood transfusion are also recorded.
Inflammatory and immune response | 7 days
  The daily highest body temperature before discharge and the values of white blood cell count, hemoglobin, C-reactive protein, prealbumin and relevant immune cytokines including IL-6, T cell count, T-helper lymphocytes (CD4+) count, T-suppressor lymphocytes (CD8+) count, natural killer (NK) cells count, B-lymphocytes count, and TNF-α from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Guoxin Li, M.D., Ph.D., Principal Investigator — Chinese Laparoscopic Gastrointestinal Surgery Study (CLASS) Group; Nanfang Hospital, Southern Medical University, China
Locations (14):
- China (14):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - The People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Wuhan Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Bethune First Hospital Jilin University, Changchun, Jilin
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Tangdu Hospital, the Fourth Military Medical University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Renji Hospital ，Shanghai Jiao Tong University School of Medicine, Shanghai

REFERENCES:
- [Background] Huscher CG, Mingoli A, Sgarzini G, Sansonetti A, Di Paola M, Recher A, Ponzano C. Laparoscopic versus open subtotal gastrectomy for distal gastric cancer: five-year results of a randomized prospective trial. Ann Surg. 2005 Feb;241(2):232-7. doi: 10.1097/01.sla.0000151892.35922.f2. PMID 15650632
- [Background] Sakuramoto S, Sasako M, Yamaguchi T, Kinoshita T, Fujii M, Nashimoto A, Furukawa H, Nakajima T, Ohashi Y, Imamura H, Higashino M, Yamamura Y, Kurita A, Arai K; ACTS-GC Group. Adjuvant chemotherapy for gastric cancer with S-1, an oral fluoropyrimidine. N Engl J Med. 2007 Nov 1;357(18):1810-20. doi: 10.1056/NEJMoa072252. PMID 17978289
- [Background] Kim HH, Hyung WJ, Cho GS, Kim MC, Han SU, Kim W, Ryu SW, Lee HJ, Song KY. Morbidity and mortality of laparoscopic gastrectomy versus open gastrectomy for gastric cancer: an interim report--a phase III multicenter, prospective, randomized Trial (KLASS Trial). Ann Surg. 2010 Mar;251(3):417-20. doi: 10.1097/SLA.0b013e3181cc8f6b. PMID 20160637
- [Background] Songun I, Putter H, Kranenbarg EM, Sasako M, van de Velde CJ. Surgical treatment of gastric cancer: 15-year follow-up results of the randomised nationwide Dutch D1D2 trial. Lancet Oncol. 2010 May;11(5):439-49. doi: 10.1016/S1470-2045(10)70070-X. Epub 2010 Apr 19. PMID 20409751
- [Derived] Wei LH, Zheng HL, Liu ZY, Du XQ, Chen CS, Xu BB, Zheng HH, Lin GT, Xie JW, Zheng CH, Wang JB, Huang CM, Li P. Preoperative visceral fat area predicts intraoperative adverse events during lymphadenectomy in laparoscopic gastrectomy for gastric cancer: a post hoc analysis. Surg Endosc. 2025 Apr;39(4):2275-2287. doi: 10.1007/s00464-025-11602-x. Epub 2025 Feb 12. PMID 39937241
- [Derived] Liu ZY, Chen QY, Zhong Q, Li P, Xie JW, Wang JB, Lin JX, Lu J, Cao LL, Lin M, Huang CM, Zheng CH. Intraoperative Adverse Events, Technical Performance, and Surgical Outcomes in Laparoscopic Radical Surgery for Gastric Cancer: A Pooled Analysis From 2 Randomized Trials. Ann Surg. 2023 Aug 1;278(2):222-229. doi: 10.1097/SLA.0000000000005727. Epub 2022 Oct 17. PMID 36250322
- [Derived] Huang C, Liu H, Hu Y, Sun Y, Su X, Cao H, Hu J, Wang K, Suo J, Tao K, He X, Wei H, Ying M, Hu W, Du X, Yu J, Zheng C, Liu F, Li Z, Zhao G, Zhang J, Chen P, Li G; Chinese Laparoscopic Gastrointestinal Surgery Study (CLASS) Group. Laparoscopic vs Open Distal Gastrectomy for Locally Advanced Gastric Cancer: Five-Year Outcomes From the CLASS-01 Randomized Clinical Trial. JAMA Surg. 2022 Jan 1;157(1):9-17. doi: 10.1001/jamasurg.2021.5104. PMID 34668963
- [Derived] Ji JF. [Chinese standard and milestone of laparoscopic surgery for gastric cancer--Comments on the publishing of "Standard Operation Procedure of Laparoscopic surgery from CLASS-01 trial"]. Zhonghua Wei Chang Wai Ke Za Zhi. 2019 Oct 25;22(10):913-915. doi: 10.3760/cma.j.issn.1671-0274.2019.10.002. Chinese. PMID 31630485
- [Derived] Yu J, Huang C, Sun Y, Su X, Cao H, Hu J, Wang K, Suo J, Tao K, He X, Wei H, Ying M, Hu W, Du X, Hu Y, Liu H, Zheng C, Li P, Xie J, Liu F, Li Z, Zhao G, Yang K, Liu C, Li H, Chen P, Ji J, Li G; Chinese Laparoscopic Gastrointestinal Surgery Study (CLASS) Group. Effect of Laparoscopic vs Open Distal Gastrectomy on 3-Year Disease-Free Survival in Patients With Locally Advanced Gastric Cancer: The CLASS-01 Randomized Clinical Trial. JAMA. 2019 May 28;321(20):1983-1992. doi: 10.1001/jama.2019.5359. PMID 31135850
- See also: Southern Medical University, China — http://www.fimmu.com/index_com.html
- See also: Nanfang Hospital, China — http://www.nfyy.com/
- See also: Chinese Anti-Cancer Association — http://www.caca.org.cn/